CLINICAL TRIAL: NCT00251849
Title: Prospective Evaluation of Rifalazil Effect On Vascular Symptoms of Intermittent Claudication and Other Endpoints in Chlamydia Seropositive Patients
Brief Title: PROVIDENCE-1: Study of Rifalazil in Chlamydia Pneumoniae Seropositive Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ActivBiotics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABI-1648-022
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2006-10

CONDITIONS: Peripheral Vascular Diseases; Intermittent Claudication
Keywords: Intermittent Claudication
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication | interventions — KRM 1648

INTERVENTIONS:
Drug: Rifalazil

SUMMARY:
The objective of this study is to determine whether rifalazil can significantly increase peak walking time (PWT) in patients with peripheral arterial disease (PAD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 40 and 80 years of age, inclusive.
* The patient has seropositive evidence of Chlamydia pneumoniae defined by immunoglobulin G antibody titers.
* The patient has a diagnosis of intermittent claudication due to PAD at screening.
* The patient's maximal effort PWT is limited only by severe claudication symptoms.
* If the patient is taking cilostazol or pentoxifylline and has been on a stable dose of the medication for at least 6 months prior to screening. Patients who have recently discontinued medications for PAD and/or intermittent claudication must "wash-out" for at least one month prior to screening.
* The patient has been on a stable dose of statin therapy for at least 6 months prior to screening.Patients who have recently discontinued statin therapy must "wash-out" for at least one month prior to screening.
* Male and female patients must agree to use an effective form of birth control throughout the study period.

Exclusion Criteria:

* The patient has critical limb ischemia as evidenced by ischemic rest pain, ulceration, or gangrene.
* The patient has had a major amputation of the leg or any other amputation that limits walking ability.
* The patient is planned for surgical/endovascular intervention for PAD during the course of the study.
* The patient has or is being treated or evaluated for tuberculosis.
* The patient has a known immunodeficient state (e.g., positive for human immunodeficiency virus) or is being treated with immunosuppressive drugs including high dose steroids or cyclosporine.
* The patient has an active infection requiring systemic or oral antibiotics.
* The patient has an uncontrolled, unstable or recently diagnosed autoimmune disease, including but not limited to systemic lupus, inflammatory bowel disease, sarcoidosis, rheumatoid arthritis, or psoriasis. Patients who develop autoimmune disease during the course of the study must be withdrawn.
* The patient's PWT is limited by symptoms other than claudication (shortness of breath, fatigue, angina, or arthritis).
* The patient has a history of alcohol abuse, illicit drug use or drug abuse or significant mental illness.
* The patient has a known or suspected allergy to the study medication(s) or class of study medication (rifamycins) to be administered.
* The patient chronically uses antibacterials or has previously received rifalazil or any rifamycin (e.g. rifampin).
* The patient has uncontrolled hypertension (resting blood pressure > 160/100 mm Hg), uncontrolled moderate to severe congestive heart failure (CHF), or uncontrolled arrhythmic disorders.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274
Dates: Start 2005-11; Study Completion 2007-12

PRIMARY OUTCOMES:
The efficacy endpoint is change from baseline in PWT
The safety endpoints are adverse event rates, rates of clinically significant laboratory abnormalities, vital signs, and physical exam abnormalities, rate of vascular death, myocardial infarction (MI), stroke, revascularization or vascular procedures

CONTACTS AND LOCATIONS:
Locations (47):
- United States (23):
  - Scottsdale Cardiovascular Research Institute, Scottsdale, Arizona
  - VA Palo Alto Health Care System, Palo Alto, California
  - Siddeg, Inc., San Diego, California
  - Apex Research Institute, Santa Ana, California
  - Radiant Research, Santa Rosa, California
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University Clinical Research, Pembrook Pines, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Rockdale Medical Research Associates, Conyers, Georgia
  - The Care Group, Indianapolis, Indiana
  - Androscoggin Cardiology Associates, Auburn, Maine
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - St. Louis University, St Louis, Missouri
  - Durham VA Medical Center, Durham, North Carolina
  - New Hope Research of Oregon, Inc., Portland, Oregon
  - Radiant Research, Philadelphia, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Black Hills Clinical Research Center, Rapid City, South Dakota
  - Hampton Roads Center for Clinical Research, Norfolk, Virginia
  - National Clinical Research, Richmond, Virginia
  - Care Foundation, Wausau, Wisconsin
- Brazil (6):
  - Hospital e Maternidade Dr. Christovao da Gama, Santo André, São Paulo
  - Centro de Ciencias Medicas e Biologicas da Pontificia Universidade, Sorocaba, São Paulo
  - Depto de Cirurgia e ortopedia, Botucatu
  - SMHS - Area Especial, Brasília
  - Hospital Pedro Ernesto, Rio de Janeiro
  - Instituto de molestias cardiovasculares, São José do Rio Preto
- Russia (18):
  - Vishnevsky Institute of Surgery, Moscow
  - Russian State Medical University, Moscow
  - Central Clinical Hospital #1, Moscow
  - City Hospital # 13, Nizhny Novgorod
  - Meshalkin Research Institute of Blood Circulation Pathology, Novosibirsk
  - Dzhanelidze Emergency Medicine Research Institutes, Saint Petersburg
  - Saint Petersburg Djanelidze Research Institute of First Aid, Saint Petersburg
  - Saint Petersburg State Medical Pediatric Academy, Saint Petersburg
  - Research Institute of Cardiology n.a. Almazov, Saint Petersburg
  - City Hospital #2, Saint Petersburg
  - City Hospital #26, Saint Petersburg
  - Saint Petersburg Pavlov Medical University, Saint Petersburg
  - Pokrovskaya Hospital, Saint Petersburg
  - City Clinical Hospital # 1, Saratov
  - Clinical Hospital #1, Smolensk
  - Tomsk Research Center, Tomsk
  - Regional Clinical Hospital, Vladimir
  - Clinical City Hospital # 25, Volgograd

REFERENCES:
- [Derived] Jaff MR, Dale RA, Creager MA, Lipicky RJ, Constant J, Campbell LA, Hiatt WR. Anti-chlamydial antibiotic therapy for symptom improvement in peripheral artery disease: prospective evaluation of rifalazil effect on vascular symptoms of intermittent claudication and other endpoints in Chlamydia pneumoniae seropositive patients (PROVIDENCE-1). Circulation. 2009 Jan 27;119(3):452-8. doi: 10.1161/CIRCULATIONAHA.108.815308. Epub 2009 Jan 12. PMID 19139383